CLINICAL TRIAL: NCT02727660
Title: A Randomized, Double-Blind, Parallel Group, Multi-Center Study to Assess the Efficacy and Safety of PT009 Compared to PT005 on COPD Exacerbations Over a 52-Week Treatment Period in Subjects With Moderate to Very Severe COPD
Brief Title: A Study to Assess the Efficacy and Safety of PT009 Compared to PT005 on COPD Exacerbations Over a 52-Week Period in Subjects With Moderate to Very Severe COPD (Sophos)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT009003
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disorder
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BFF MDI (PT009) 320/9.6 μg (Experimental): Budesonide and Formoterol Fumarate Inhalation Aerosol - 160/4.8 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: BFF MDI (PT009) 320/9.6 μg
- BFF MDI (PT009) 160/9.6 μg (Experimental): Budesonide and Formoterol Fumarate Inhalation Aerosol - 80/4.8 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: BFF MDI (PT009) 160/9.6 μg
- FF MDI (PT005) 9.6 μg (Experimental): Formoterol Fumarate Inhalation Aerosol - 4.8 μg per actuation MDI/120 inhalations Taken as 2 inhalations BID
  Interventions: Drug: FF MDI (PT005) 9.6 μg

INTERVENTIONS:
Drug: BFF MDI (PT009) 320/9.6 μg — Blinded Treatment
  Other Names: Budesonide and Formoterol Fumarate Inhalation Aerosol
  Arms: BFF MDI (PT009) 320/9.6 μg
Drug: BFF MDI (PT009) 160/9.6 μg — Blinded Treatment
  Other Names: Budesonide and Formoterol Fumarate Inhalation Aerosol
  Arms: BFF MDI (PT009) 160/9.6 μg
Drug: FF MDI (PT005) 9.6 μg — Blinded Treatment
  Other Names: Formoterol Fumarate Inhalation
  Arms: FF MDI (PT005) 9.6 μg

SUMMARY:
This is a Phase III randomized, double-blind, parallel group, multi-center, 52-week COPD exacerbation and lung function study with PT009 320/9.6 μg, PT009 160/9.6 μg and PT005 9.6 μg, all administered BID.

DETAILED DESCRIPTION:
This is a Phase III randomized, double-blind, parallel group, multi-center, 52-week COPD exacerbation and lung function study. Subjects will undergo a 1- to 4-week Screening Period. Subjects who successfully complete the Screening Period will be randomized to one of the following three treatment groups: PT009 320/9.6 μg, PT009 160/9.6 μg and PT005 9.6 μg, all administered BID. Following randomization, subjects will enter the Treatment Period and undergo additional treatment visits over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Give their signed written informed consent to participate
2. At least 40 years of age and no older than 80 years of age
3. COPD patients who are symptomatic
4. Must be receiving one or more inhaled bronchodilators as maintenance therapy
5. Must have a documented history of COPD exacerbations

Exclusion Criteria:

1. Current diagnosis of asthma
2. COPD due to α1-Antitrypsin Deficiency
3. Known active tuberculosis, lung cancer, cystic fibrosis, and significant bronchiectasis, Pulmonary resection or Lung Volume Reduction Surgery during the past 6 months.
4. Long-term-oxygen therapy (≥ 15 hours a day).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1876 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (240):
- United States (110):
  - Research Site, Dothan, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Flagstaff, Arizona
  - Research Site, Costa Mesa, California
  - Research Site, Gold River, California
  - Research Site, Lincoln, California
  - Research Site, Long Beach, California
  - Research Site, Palo Alto, California
  - Research Site, San Diego, California
  - Research Site, Upland, California
  - Research Site, Yorba Linda, California
  - Research Site, Boulder, Colorado
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Chiefland, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Lehigh Acres, Florida
  - Research Site, Merritt Island, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Dacula, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Aurora, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Olathe, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Hazard, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Biddeford, Maine
  - Research Site, Rochester, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Toms River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Gastonia, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Cumberland, Rhode Island
  - Research Site, East Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Lancaster, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Smyrna, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Baytown, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Lufkin, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, Port Arthur, Texas
  - Research Site, Sherman, Texas
  - Research Site, Spring, Texas
  - Research Site, Waco, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Manassas, Virginia
  - Research Site, Everett, Washington
  - Research Site, Renton, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (15):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonomade Buenos Aires
  - Research Site, Ciudad Autónoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Concepción del Uruguay
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Austria (4):
  - Research Site, Bludenz
  - Research Site, Feldbach
  - Research Site, Hallein
  - Research Site, Linz
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Erpent
  - Research Site, Gilly
  - Research Site, Jambes
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (8):
  - Research Site, Botucatu
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
  - Research Site, Sorocaba
  - Research Site, Uberlândia
  - Research Site, Vitória
- Canada (5):
  - Research Site, Ajax, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (4):
  - Research Site, Curicó
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Talcahuano
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, København NV
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Silkeborg
- Germany (7):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Cottbus
  - Research Site, Frankfurt
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Rodgau-Dudenhofen
- Italy (12):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Ferrara
  - Research Site, Legnago
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Riccione
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Sassari
- Mexico (7):
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Minatitlán
  - Research Site, Monterrey
  - Research Site, Sonora
  - Research Site, Villahermosa
- Norway (6):
  - Research Site, Arendal
  - Research Site, Hønefoss
  - Research Site, Kråkeroy
  - Research Site, Stavanger
  - Research Site, Svelvik
  - Research Site, Trondheim
- Peru (4):
  - Research Site, Chancay
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Piura
- Puerto Rico (2):
  - Research Site, Ponce
  - Research Site, San Juan
- Russia (10):
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, StPetersburg
  - Research Site, Ulyanovsk
  - Research Site, Yekaterinburg
- South Africa (9):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, KwaDukuza
  - Research Site, Lenasia Ext8
  - Research Site, Mowbray
  - Research Site, Parow
  - Research Site, Pretoria
- Spain (12):
  - Research Site, Alicante
  - Research Site, Alzira (Valencia)
  - Research Site, Benalmádena (Málaga)
  - Research Site, Cáceres
  - Research Site, Jerez de la Frontera
  - Research Site, Laredo
  - Research Site, Loja (Granada)
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Sagunto(Valencia)
  - Research Site, Sant Boi de Llobregat
- Sweden (4):
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala
- United Kingdom (7):
  - Research Site, Bradford
  - Research Site, Chertsey
  - Research Site, Chester
  - Research Site, Doncaster
  - Research Site, Lancaster
  - Research Site, Sheffield
  - Research Site, Wishaw

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4138&filename=PT009003_Protocol_Redacted_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4138&filename=PT009003_SAP_Redacted_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study screened subjects at 292 study centers in 18 countries and randomized subjects at 259 study centers, from April 2016 to April 2018.
Pre-assignment Details: Subjects were randomized in a 1:1:1 ratio to BFF MDI 320/9.6 μg, BFF MDI 160/9.6 μg, and FF MDI 9.6 μg treatment groups
Groups:
- BFF MDI 320/9.6 ug: Budesonide Formoterol Fumarate Metered dose inhalation 320/9.6 ug
- BFF MDI 160/9.6 ug: Budesonide Formoterol Fumarate Metered dose inhalation 160/9.6 ug
- FF MDI 9.6 ug: Formoterol Fumarate Metered dose inhalation 9.6 ug
Period: Overall Study
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
Started (mITT Population) | 619 | 617 | 607
Completed (Completed Study Treatment) | 503 | 501 | 442
Not Completed | 116 | 116 | 165
Not completed — Lack of Efficacy | 40 | 40 | 70
Not completed — Adverse Event | 28 | 21 | 32
Not completed — Withdrawal by Subject | 26 | 25 | 30
Not completed — Physician Decision | 3 | 8 | 14
Not completed — Lost to Follow-up | 5 | 9 | 8
Not completed — Protocol Violation | 7 | 5 | 5
Not completed — Protocol Specified Disc. Criteria | 5 | 5 | 2
Not completed — Administrative Reasons | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) Population is defined as all subjects who were randomized to treatment (presented here). The Modified Intent-To-Treat (mITT) Population, a subset of the ITT Population, is defined as all subjects with post-randomization data obtained prior to d/c from treatment. The mITT Population was used for all efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug | Total
Number analyzed (Participants) | 629 | 630 | 617 | 1876
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: mITT Population
  Years
    number analyzed (Participants) | 619 | 617 | 607 | 1843
    (all) | 65.3 (8.1) | 64.5 (8.4) | 64.8 (8.5) | 64.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 619 | 617 | 607 | 1843
    Female | 252 | 272 | 268 | 792
    Male | 367 | 345 | 339 | 1051
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 619 | 617 | 607 | 1843
    Hispanic or Latino | 190 | 200 | 190 | 580
    Not Hispanic or Latino | 423 | 414 | 412 | 1249
    Unknown or Not Reported | 6 | 3 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 619 | 617 | 607 | 1843
    American Indian or Alaska Native | 26 | 18 | 24 | 68
    Asian | 1 | 7 | 4 | 12
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Black or African American | 30 | 22 | 29 | 81
    White | 514 | 516 | 504 | 1534
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 47 | 54 | 46 | 147

OUTCOME MEASURES:

1. Primary Outcome: Morning Pre-dose Trough FEV1
Description: Morning pre-dose trough FEV1 (Forced Expiratory Volume in one second) at week 12
Time Frame: at Week 12
Population: mITT Population Only subjects who had morning pre-dose trough FEV1 measured at the week 12 visit are included in the "at Week 12" timepoint
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 542 | 540 | 501
Liter | 0.072 [0.053 to 0.090] | 0.069 [0.051 to 0.087] | 0.037 [0.018 to 0.056]

2. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation
Description: Time to first moderate or severe COPD (Chronic Obstructive Pulmonary Disease) exacerbation over 52 weeks
Time Frame: over 52 weeks
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects with Exacerbation
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 619 | 617 | 607
Percentage of Subjects with Exacerbation
  Percent of Subjects Exacerbated within 12 Weeks | 19.2 [16.2 to 22.6] | 19.3 [16.3 to 22.7] | 24.8 [21.5 to 28.6]
  Percent of Subjects Exacerbated within 24 Weeks | 31.2 [27.5 to 35.4] | 32.9 [29.1 to 37.1] | 35.1 [31.3 to 39.4]
  Percent of Subjects Exacerbated within 36 Weeks | 41.0 [36.5 to 45.9] | 41.3 [36.9 to 46.0] | 46.2 [41.5 to 51.2]
  Percent of Subjects Exacerbated within 52 Weeks | 50.1 [44.4 to 56.0] | 48.6 [43.1 to 54.4] | 54.8 [49.0 to 60.7]

3. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin HFA Use
Description: Change from baseline in average daily rescue Ventolin HFA use over 12 weeks
Time Frame: over 12 weeks
Population: mITT Population Only subjects who had rescue Ventolin HFA doses recorded over the 12 week period are included in the "over 12 Weeks" timepoint
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs per day
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 612 | 610 | 599
Puffs per day | -0.9 [-1.1 to -0.7] | -0.9 [-1.1 to -0.7] | -0.6 [-0.8 to -0.4]

4. Secondary Outcome: Percentage of Subjects Achieving an MCID (Minimal Clinically Important Difference) of 4 Units or More in Saint George's Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ (St. George's Respiratory Questionnaire) is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of BFF MDI on health-related quality of life as compared to FF MDI in subjects with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. A decrease from baseline in SGRQ total score of 4 units or more is considered a clinically meaningful improvement in quality of life.
Time Frame: at Week 12
Population: mITT Population
Measure: Number; unit: Percentage of Subjects
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
Number analyzed (Participants) | 619 | 617 | 607
Percentage of Subjects | 52 | 54 | 44

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug.
Description: Serious Adverse Events were collected from the time the subject signed informed consent throughout the treatment period and up to approximately 52 weeks, which includes screening and follow up (14 days after last dose of study drug).
Arm/Group | BFF MDI 320/9.6 ug | BFF MDI 160/9.6 ug | FF MDI 9.6 ug
All-Cause Mortality (participants affected / at risk) | 3/619 | 4/617 | 8/607
Serious Adverse Events (participants affected / at risk) | 60/619 | 78/617 | 83/607
Other Adverse Events (participants affected / at risk) | 266/619 | 279/617 | 268/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 ug (N=619) | BFF MDI 160/9.6 ug (N=617) | FF MDI 9.6 ug (N=607)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 30 (33) | 50 (65)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 12 (12) | 9 (9)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hydrocele male infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pnuemonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonae (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type II diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 320/9.6 ug (N=619) | BFF MDI 160/9.6 ug (N=617) | FF MDI 9.6 ug (N=607)
Nasopharyngitis (Infections and infestations) | 41 (53) | 53 (61) | 36 (43)
Upper respiratory tract infection (Infections and infestations) | 28 (29) | 14 (18) | 24 (28)
Pneumonia (Infections and infestations) | 14 (14) | 19 (20) | 15 (15)
Influenza (Infections and infestations) | 15 (15) | 19 (20) | 10 (10)
Bronchitis (Infections and infestations) | 11 (11) | 13 (15) | 10 (14)
Sinusitis (Infections and infestations) | 9 (9) | 9 (11) | 13 (13)
Acute sinusitis (Infections and infestations) | 2 (2) | 6 (10) | 12 (17)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 30 (33) | 50 (65)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 16 (19) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 10 (11) | 10 (11)
Headache (Nervous system disorders) | 16 (24) | 19 (24) | 18 (20)
Hypertension (Vascular disorders) | 15 (15) | 15 (15) | 14 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (21) | 17 (17) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 15 (17) | 9 (9)
Oral candidiasis (Infections and infestations) | 13 (16) | 6 (7) | 7 (8)
Urinary tract infection (Infections and infestations) | 10 (12) | 18 (20) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02727660/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT02727660/SAP_001.pdf